CLINICAL TRIAL: NCT03798730
Title: Investigation of the Perception of Protein Fortified Foods and Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Lisa Methven, Professor in Food and Sensory Science, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UREC 18/46
Record Dates: First submitted 2018-12-18; First posted 2019-01-10 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Individual Difference; Food Sensitivity; Food Preferences
Keywords: Older Adults; Oral Nutritional Supplements; Saliva Flow; Mucoadhesion; Mouthdrying
MeSH Terms: conditions — Food Intolerance; Food Preferences

STUDY DESIGN:
Intervention Model Description: This study involves both a crossover design where each participant tastes both the control product (not fortified) and the protein fortified product with an appropriate break between the two sessions. It is also both a within and between groups design as the responses from the older participants will be compared to the younger participants. The study will be conducted single blind as it not feasible to blind the researcher. Each participant will attend 3 study visits and all foods will be presented with random blinding codes.
Who Masked: Participant
Masking Description: All samples provided to the participant are labelled with 3 digit random codes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solid Model (Experimental): 1. Cake
     -Control Vanilla Cake and Protein Fortified Vanilla Cake
  2. Biscuit -Control Lemon Biscuit and Protein Fortified Lemon Biscuit
  Interventions: Behavioral: Solid Model
- Liquid Model (Experimental): Whey Protein Beverages
  * Native sample (protein unheated)
  * Denatured whey protein (protein heated to denature)
  Interventions: Behavioral: Liquid Model

INTERVENTIONS:
Behavioral: Solid Model — Cake and biscuit will be used, with the amount of protein varied to study the effect on perception of the products (using sensory methods of rating drying and discrimination tests "which is the stronger in drying")
  Arms: Solid Model
Behavioral: Liquid Model — Intervention Description: To study the effect of protein denaturation on perception of whey protein beverages using sensory methods (rating drying as well as discrimination tests "which is the stronger in drying"). Measuring mucoadhesion via protein content remaining in saliva following swallowing of whey protein beverages.
  Arms: Liquid Model

SUMMARY:
This study aims to investigate whether protein fortification of foods and beverages causes mouthdrying and mucoadhesion and whether this is influenced by age and saliva flow.

DETAILED DESCRIPTION:
1. To investigate, by using protein fortified foods and beverages, whether mucoadhesion to the oral cavity is greater for older adults compared to younger adults and determine whether it is related to salivary flow rate.
2. To determine whether protein fortification of foods and beverages causes mouthdrying and whether perception and acceptance are influenced by age and individual differences in saliva flow.

These aims will be investigated using two different models: a liquid model using whey protein and a solid model using protein fortified biscuits and cakes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years or over 65 years
* Self reported as healthy (no specific disease states)

Exclusion Criteria:

* Cognitively impaired
* Allergies or intolerances that include coeliac disease, lactose or gluten intolerance
* Diabetic
* Had oral surgery
* Had stroke
* Smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Saliva sample to examine change over time of protein remaining in mouth (Mucoadhesion) | Saliva collection at 4 timepoints post swallowing of each sample (15s, 30s, 60s, 120s) at study visits two and three, reported at 1 year.
  Participants drink whey protein beverages (unheated and heated protein) then after different time points post swallowing (15 seconds to 5 minutes) expectorated saliva is collected to analyse protein for the extent of mucoadhesion)

SECONDARY OUTCOMES:
Mouthdrying from cake | At one time point (visit 3) reported at 1 year.
  Perceived mouth drying from protein fortified vanilla cake and control vanilla cake using data from sensory methods (rating drying as well as discrimination tests "which is the stronger in drying")
Mouthdrying from biscuits | At one time point (visit 2) reported at 1 year.
  Perceived mouth drying from protein fortified lemon biscuits and control lemon biscuit using data from sensory methods (rating drying as well as discrimination tests "which is the stronger in drying")
Mouthdrying from whey protein | At one time point (visit 1) reported at 1 year.
  Perceived mouth drying from whey protein beverages (unheated and heated whey protein) using data from sensory methods (rating drying as well as discrimination tests "which is the stronger in drying")
Saliva Collection | Reported at 1 year (Unstimulated saliva flow taken at the start of every study visit. Stimulated saliva flow taken at the start of study visit one.)
  Salivary flow rates from unstimulated and stimulated saliva samples.
Questionnaire | At one time point (visit 1) reported at 1 year.
  Dental status and mouth behaviour categorisation via a questionnaire. Category data (ie participants check boxes that apply). The dental status questionnaire is adapted from the WHO oral health questionnaire, it indicates where a participant has poor dental status. The mouth behaviour questionnaire is a validated questionnaire (JMBM, trademarked), we are investigating whether it relates to perception of protein fortified foods.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Bull SP, Hong Y, Khutoryanskiy VV, Parker JK, Faka M, Methven L. Whey protein mouth drying influenced by thermal denaturation. Food Qual Prefer. 2017 Mar;56(Pt B):233-240. doi: 10.1016/j.foodqual.2016.03.008. PMID 28260840
- [Background] Withers CA, Cook MT, Methven L, Gosney MA, Khutoryanskiy VV. Investigation of milk proteins binding to the oral mucosa. Food Funct. 2013 Nov;4(11):1668-74. doi: 10.1039/c3fo60291e. PMID 24092277
- [Background] Affoo RH, Foley N, Garrick R, Siqueira WL, Martin RE. Meta-Analysis of Salivary Flow Rates in Young and Older Adults. J Am Geriatr Soc. 2015 Oct;63(10):2142-51. doi: 10.1111/jgs.13652. Epub 2015 Oct 12. PMID 26456531
- [Background] Gosney M. Are we wasting our money on food supplements in elder care wards? J Adv Nurs. 2003 Aug;43(3):275-80. doi: 10.1046/j.1365-2648.2003.02710.x. PMID 12859786
- [Background] Kennedy O, Law C, Methven L, Mottram D, Gosney M. Investigating age-related changes in taste and affects on sensory perceptions of oral nutritional supplements. Age Ageing. 2010 Nov;39(6):733-8. doi: 10.1093/ageing/afq104. Epub 2010 Sep 22. PMID 20861088
- [Background] Withers CA, Lewis MJ, Gosney MA, Methven L. Potential sources of mouth drying in beverages fortified with dairy proteins: A comparison of casein- and whey-rich ingredients. J Dairy Sci. 2014 Mar;97(3):1233-47. doi: 10.3168/jds.2013-7273. Epub 2014 Jan 17. PMID 24440265